CLINICAL TRIAL: NCT03788993
Title: A Pragmatic Effectiveness Randomized Controlled Trial of Duration of Psychiatric Hospitalization in a Trans-diagnostic Sample of Patients With Acute Mental Illness Admitted to a Ward With Either Blue Depleted Evening Lighting or Normal Lighting Conditions.
Brief Title: Testing the Effectiveness of an Evening Blue-depleted Light Environment in an Acute Psychiatric Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/916
Record Dates: First submitted 2018-12-20; First posted 2018-12-28 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-02

CONDITIONS: Mental Disorder
Keywords: Phototherapy; Hospitals, psychiatric; Emergency Services, Psychiatric
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: This is a single-centre, unblinded, two-arm, parallel-group, pragmatic effectiveness RCT of differences in the mean duration of acute psychiatric hospitalization in days for individuals exposed to experimental lighting compared with normal lighting conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue-depleted evening light condition (Experimental)
  Interventions: Other: Blue-depleted evening light condition
- Normal light condition (Active Comparator)
  Interventions: Other: Normal light condition

INTERVENTIONS:
Other: Blue-depleted evening light condition — A 20-bedded ward with tunable light emitting diode (LED) lamps. At 18:00h the lighting undergoes a 30-minute transition during which the green and blue LEDs are dimmed to produce blue-depleted amber colored lighting. At 06:50h a new 10-minute transition changes the light color to ordinary indoor lighting. From 07:00h to 18:00h, there is ordinary indoor lighting (3000K colour temperature). The light intensity is dimmed to 20% of the maximum from 23:00h to 6:50h.
  Blue-blocking window filters are deployed also in the evening. All TV sets have permanent blue-blocking filters and individuals are provided with blue-blocking screens that can be attached to the front of personal electronic devices. If the patients leave the blue-depleted unit after 18:30 they are offered blue-blocking glasses to wear. The light spectrum in the ward was assessed prior to commencing the RCT and is well-matched to what has been shown in laboratory settings to minimally suppress melatonin.
  Arms: Blue-depleted evening light condition
Other: Normal light condition — The other half of the unit (20 patient rooms and their corresponding bathrooms and common areas) have ordinary indoor light installed (Glamox, Norway). This has a 3000K color temperature. The light is dimmed to 20% of max in the night, similar to the blue-depleted condition.
  The light in the normal light condition and the blue-depleted light condition have similar levels of photopic lux throughout the 24h cycle, but different levels of melanopic lux between 1830h and 0700h.
  Arms: Normal light condition

SUMMARY:
There is increasing recognition of the need to stabilize sleep-wake cycles in individuals with major mental disorders. As such, clinicians and researchers advocate for the use of interventions targeted at sleep and circadian dysrhythmias as an adjunct to the standard treatments offered for acute illness episodes of a broad range of diagnoses. To determine the trans-diagnostic generalizability of chronotherapy, the investigators will explore the benefits of admitting individuals with major mental disorders to an acute psychiatric inpatient unit where changes in light exposure are integrated into the therapeutic environment.

A two-arm pragmatic effectiveness randomized controlled treatment trial, where individuals admitted for inpatient psychiatric care will be allocated to a ward with blue depleted evening light or to a ward with the same layout and facilities but lacking the new lighting technology. The trial will test whether the experimental lighting conditions offer any additional benefits beyond those associated with usual treatment in an acute psychiatric inpatient unit.

The main objectives are to examine any differences between groups in the mean duration of hospitalization in days. Additional analyses will compare groups differences in sleep, functioning, symptoms, medication usage, and side-effects and whether length of stay is associated with stability of sleep-wake cycles and circadian rhythms. Given this unique research opportunity, ancillary investigations will determine any benefits according to diagnostic subgroups and potential drawbacks such as any adverse effects on the well-being of professionals working across both wards.

DETAILED DESCRIPTION:
In recent decades there has been increased attention to the impact of disturbed sleep on general health. For example, sleep-wake cycle abnormalities linked with circadian dysrhythmias are associated with physical disorders such as diabetes, metabolic abnormalities, obesity, impaired functioning of the immune system, and a greater risk of cancer. Given that light is a central zeitgeber of the circadian system, this had led to some researchers exploring the benefits of photo- or chrono-therapies for selected medical illnesses, especially in those individuals who have a concurrent comorbid mental disorder. The latter is noteworthy as sleep problems are uniquely important in the field of mental health. For instance, sleep abnormalities may be prodromal symptoms that precede the onset of a first episode of a major mental disorder, sleep-wake cycle disruptions are criterion symptoms of unipolar and bipolar disorders and circadian dysrhythmias may exacerbate suicidal behaviours. In addition, research demonstrates that day-to-day variability in the sleep-wake cycle is associated with longer duration of admission to an acute psychiatric inpatient unit and frequency of aggressive behavior and violent incidents. Lastly, and importantly, sleep problems are often the last clinical symptoms to resolve during recovery from an acute episode of a mood or psychotic disorder. Overall, experimental and clinical research emphasize the reciprocal relationship between sleep-wake disruptions and mental disorders showing that they perpetuate and exacerbate each other and that improved sleep is associated with improvements in mental state.

The observations noted above have increased awareness of the need to stabilize sleep-wake cycles in individuals with major mental disorders and highlighted the importance of incorporating therapeutic interventions targeted at circadian dysrhythmias as an adjunct to other treatments offered for acute illness episodes. Psychological and pharmacological interventions are efficacious approaches for sleep-wake cycle disturbances in adults without comorbid mental disorders. However, their use in individuals with an acute exacerbation of a major mental illness can be problematic, including attenuation of the benefit-to-risk ratio for therapies or contra-indications to the use of some medications. Partly as a response to these concerns, but also because of new research on circadian rhythms, attention has shifted to the potential role of chronotherapeutic interventions based on controlled exposures to environmental stimuli that act on biological rhythms. These strategies initially focused on e.g. bright light therapy for seasonal affective disorders and for some sub-types of depression; but more recently they have been extended to e.g. dark therapy (spending 14 hours in darkness per day) or the use of blue blocking glasses in for patients who are hospitalized for the treatment of acute mania. To date, clinical trials of all these interventions have been targeted at small and/or homogeneous samples with a specified sleep or mood disorder (e.g. delayed sleep phase syndrome or bipolar depression, etc.) and have required the study participants to adhere to a protocol for the repeated use of equipment at specified times of the day (sitting by a lamp, resting in forced darkness or wearing glasses, etc.).

The above represent interesting treatment advances. However, given the prevalence of sleep-wake cycle disturbances in individuals with mental disorders, it is logical to extend trials of the use of these types of interventions to broader trans-diagnostic populations. Furthermore, to enhance the generalizability of interventions, it would be helpful to avoid giving personal responsibility for following protocols regarding exposure to different intensities or spectra of light to individuals who are acutely unwell. A pragmatic alternative is to create a therapeutic environment for patients with major mental disorders where changes in light exposure are regulated automatically and where programable lighting conditions form an integral part of a hospital unit. This is an intriguing option as little consideration has been given to how contemporary technology might be employed to augment any benefits of acute treatment in an inpatient facility. Historically, acute psychiatric admission units have offered asylum and a place of safety, and it is assumed that ward routines and structured activities may reduce arousal, regularize sleep-wake cycle patterns and improve confidence and self-esteem, etc. However, the focus is primarily on physical and pharmacological treatments that reduce symptoms and suicidality, enhance social functioning and sufficiently improves the individuals mental state to allow a timely return to outpatient or community care. Less attention has been given to the creation of a state-of-the-art inpatient milieu.

The investigators have been involved in the planning and design of a newly-built psychiatric unit and this process has allowed the investigators to consider how the inpatient environment might be modified to try to enhance recovery from acute illness. The unit comprises of two wards: one ward incorporates state-of-the-art lighting technology while the other ward has an identical layout and facilities but has normal lighting conditions. This unit offers a unique opportunity to explore how exposure to different lighting conditions may modify sleep-wake cycles and how any changes may impact on the clinical and functional outcomes of individuals experiencing an acute episode of a severe mental disorder that requires inpatient care. The findings could influence the future design of hospital units offering care to patients with mental or physical disorders.

The investigators aim to recruit 400 individuals who give written informed consent to participate in a two-arm pragmatic effectiveness randomized controlled clinical treatment trial (RCT). However, based on projected admission rates, the investigators believe that this sample size is at the lower limit of the estimated study population as they are permitted to continue recruitment for at least six consecutive months.

Eligible individuals will be allocated to a ward with a lighting system that produces an environment with blue depleted evening light or to a ward with the same layout and facilities but lacking the new lighting technology. The trial will test whether the environment with programmable lighting conditions offers any additional benefits beyond those associated with usual treatment in an acute psychiatric inpatient unit. The main objectives are to examine if there are any differences between groups in the mean duration of hospitalization. In addition, the investigators will explore whether level of functioning, day-to-day symptom ratings, episodes of suicidality or aggressive behavior, medication usage, and self-reported side-effects differ between groups and whether shorter duration of admission is associated with greater stability of sleep-wake cycles and circadian rhythms.

Given that this trail takes place in a unique setting, the investigators will undertake several ancillary investigations to determine the range of benefits or adverse effects for subpopulations of patients (e.g. different diagnostic subgroups) and examine any potential benefits or drawbacks to the use of this new lighting system, including actigraphic recordings of sleep-wake patterns of nurses and any self-reported effects on well-being that are recorded by professionals who experience working in both wards.

Update March 8th, 2019

As noted in the original protocol, we aimed to recruit a minimum of 400 individuals who give written informed consent to participate in a two-arm pragmatic effectiveness randomized controlled clinical treatment trial (RCT), with the expectation that we would actually include about 200-250 individuals per group. This recruitment target takes into account 'failure to complete randomization' (i.e. the patient is randomized to a specified lighting condition, but is not admitted to the bed in the ward with the allocated lighting condition; this may occur for a number of reasons that were listed in the original protocol) and the delayed consent procedure (we note that the delay between randomization and consent is, on average, about 14 days).

The recruitment period was about 6 months (Oct 23th 2018 until April 12th 2019), but we set a limit on randomization to March 31st and for obtaining delayed consent of April 12th. This time frame was selected as it corresponds to the winter period in this region of Norway. After March 31st, daylight saving time changes and also we experience very different environmental light exposure (long days, short nights, etc). This is relevant as it means that any extension to the recruitment period needs to be delayed until the environmental light exposure matches that experienced by individuals who entered the RCT at the start of recruitment. As such, we agreed (in advance of starting the RCT) with the ethics committee and trial steering group, that should we fall short of the target sample size after six months or recruitment, then the recruitment process would be suspended and would be re-opened in October 2019 (when the environmental light exposure would be the same as during the original winter recruitment period).

Although our projected randomization rate is as expected (and we have randomized >600 individuals by month 4-5 of the study), two issues have arisen with completion of randomization. The first was totally unpredictable, namely that a regional electricity power failure meant that we could not properly randomize admissions for a 72-hour weekend period (during with >15 admissions occurred). After discussion, it was agreed that the manual system of randomization that was introduced over that weekend could not be regarded as equivalent to the automated system, so these cases were immediately excluded from the RCT sample. Second, the bed occupancy rate in January and February has been running at about 100%, meaning that many randomizations cannot be completed (i.e. the patient is randomized but cannot then be admitted to the lighting condition to which they were allocated).

We undertook modelling of the projected number of randomizations that would be completed (i.e. admitted to the lighting condition allocated at randomization) and have given written informed consent by April 12th. the projected admission rates, we believe that this sample size is at the lower limit of the estimated study population (as we are permitted to continue recruitment for at least six consecutive months). We modelled the best- and worst-case scenario. The best-case scenario suggested we would achieve the target sample by April 12th (>400), but the worst-case scenario suggested we may only have randomized, completed correct allocation and obtained the delayed consent in about 350-360 cases.

Given the above, and the pre-trial agreement that recruitment could be suspended and re-opened in October 2019, this is course of action we have taken. As we do not break the codes for randomization (completed as allocated or failed) or match these to which individuals have given consent (via the deferred procedure), we cannot know the exact number of trial participants we need to recruit in October. However, the original protocol stated we would recruit 400-500 participants. With this in mind, we will re-open randomization for six weeks, starting October 2019, and close the consent procedure by the end of November 2019.

Added October 7t,h 2021:

The Statistical Analytical Plan (SAP) has been written before anyone have performed any analyses on data from the trial. Analyses of the data from the trial will start one week after the SAP has been uploaded to https://register.clinicaltrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18 years or older
* Admitted to the acute inpatient unit at St. Olavs University Hospital, Department Østmarka, Trondheim, Norway during the inclusion period for the study.
* Any patients who are re-admitted during the inclusion period for the study are eligible for re-randomization.

Exclusion Criteria:

Post-randomization, there are four potential reasons for exclusion from the RCT:

* Lack of availability of rooms (as allocated at randomization): acute wards operate at high levels of bed occupancy, so on some occasions there will be no rooms available in the ward to which the individual is allocated (i.e. the randomization process cannot be completed).
* Clinical imperative: on some occasions senior medical or nursing professionals may decide that it is clinically inappropriate to admit an individual to a vacant room in the ward to which they are randomized. The most frequent reasons for this to occur are clinical concerns about (a) how this admission would affect the case mix within the ward (e.g. it may be inappropriate to locate all the patients with an acute episode of mania in one ward, etc.) and/or (b) completing the randomization process may compromise the safety, care and treatment of current inpatients or of the individual being admitted (e.g. it may not be possible to provide the appropriate staff-to-patient ratio required for optimal treatment if all individuals with higher levels of need are located in one ward, etc.).
* The individual is unwilling to give written informed consent at any time during their admission (when approached according to the deferred consent procedure) or is unable to give informed consent for the duration of the study (i.e. they remain persistently and severely ill and/or lack mental capacity).
* The consent procedure was incomplete: an individual may be discharged early or have an unplanned discharge (e.g. discharge against medical advice) which may mean they were not approached about study participation or they had only given verbal, but not written consent.

Withdrawal criteria:

As randomization occurs at the point of admission, all exclusions de facto occur post-randomization, so the criteria described above represent the main reasons for study withdrawal.

Additional withdrawal criteria:

* A patient will be withdrawn from the study if they are absent for >24 hours from the ward to which they randomized (e.g. they may be transferred to a medical ward for several days; the patient may request or the clinicians instigate transfer to another ward; medical or nursing staff may decide the patient should be transferred to the other ward at the unit because of patient need, case mix or staffing issues, etc.).
* An individual can decline to participate at any stage of the study and/or a mental health professional can recommend withdrawal of an inpatient from the RCT if they have any clinical concerns regarding an individuals' participation (e.g. if there is a belief that the patient has experienced an adverse event associated with exposure to the blue-depleted light). In all instances a record will be kept of reasons for withdrawal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Duration of admission | Recorded at the date of discharge (range from 0 to about 150 days).
  The primary outcome measure will be mean duration of admission per individual. The date and time of admission and of discharge will be extracted from the electronic records for the Intention To Treat (ITT) analyses. For the per-protocol analyses discharge will be the date and time the patient left the light environment the patient was randomized to and was subsequently away from the unit for more than 24 hours.

SECONDARY OUTCOMES:
Total Sleep Time | Daily throughout the admission (range form 0 to about 150 days).
  Individual sleep and activity patterns will be assessed using de-identified data collected via radar (Xethru sensors) installed in each room and the en suite bathroom. The sensor is a low-powered ultra-wideband radar that allows contact-free assessment sleep patterns and wakefulness with high accuracy compared to polysomnographic (PSG) recordings.
  Employing best available scoring algorithms, raw data from daily recordings will be used to estimate total sleep time.
Bed time | Recorded daily throughout the admission (range form 0 to about 150 days).
  Individual sleep and activity patterns will be assessed using de-identified data collected via radar (Xethru sensors) installed in each room and the en suite bathroom. The sensor is a low-powered ultra-wideband radar that allows contact-free assessment sleep patterns and wakefulness with high accuracy compared to polysomnographic (PSG) recordings.
  Employing best available scoring algorithms, raw data from daily recordings will be used to estimate the time the patients went to bed (bed time).
Sleep onset | Recorded daily throughout the admission (range form 0 to about 150 days).
  Individual sleep and activity patterns will be assessed using de-identified data collected via radar (Xethru sensors) installed in each room and the en suite bathroom. The sensor is a low-powered ultra-wideband radar that allows contact-free assessment sleep patterns and wakefulness with high accuracy compared to polysomnographic (PSG) recordings.
  Employing best available scoring algorithms, raw data from daily recordings will be used to estimate the time for sleep onset.
Nocturnal awakenings | Recorded daily throughout the admission (range form 0 to about 150 days).
  Individual sleep and activity patterns will be assessed using de-identified data collected via radar (Xethru sensors) installed in each room and the en suite bathroom. The sensor is a low-powered ultra-wideband radar that allows contact-free assessment sleep patterns and wakefulness with high accuracy compared to polysomnographic (PSG) recordings.
  Employing best available scoring algorithms, raw data from daily recordings will be used to estimate number of nocturnal awakenings.
Wake after sleep onset | Recorded daily throughout the admission (range form 0 to about 150 days).
  Individual sleep and activity patterns will be assessed using de-identified data collected via radar (Xethru sensors) installed in each room and the en suite bathroom. The sensor is a low-powered ultra-wideband radar that allows contact-free assessment sleep patterns and wakefulness with high accuracy compared to polysomnographic (PSG) recordings.
  Employing best available scoring algorithms, raw data from daily recordings will be used to estimate the time a patient is awake after initial sleep onset.
Sleep offset | Recorded daily throughout the admission (range form 0 to about 150 days).
  Individual sleep and activity patterns will be assessed using de-identified data collected via radar (Xethru sensors) installed in each room and the en suite bathroom. The sensor is a low-powered ultra-wideband radar that allows contact-free assessment sleep patterns and wakefulness with high accuracy compared to polysomnographic (PSG) recordings.
  Employing best available scoring algorithms, raw data from daily recordings will be used to estimate the time of final awakening called sleep offset.
Level of clinical improvement | Recorded daily throughout admission and at the date of discharge (range from 0 to about 150 days).
  Clinical Global Impression, Improvement subscale (CGI-I): The investigators use the Improved version of the Clinical Global Improvement Scale (iCGI-I).28 Scores capture change over time with ratings ranging from -6 (maximum deterioration) to +6 (ideal improvement). The iCGI-I is used (a) to monitor day-to-day changes in mental state and functioning, and (b) to record overall change from admission to discharge.
Level of illness severity | First 0-24 hours of admission, last 24 hours of admission
  Clinical Global Impression, Severity subscale (CGI-S): The CGI-S is a likert scale ranging from 1 (Normal, not at all ill) to 7 (Among the most extremely ill patients). These CGI-S ratings are benchmarked relative the total inpatient population (i.e. not according to diagnostic subgroups). It is scored on two occasions only: the morning after admission to the unit (based on observations for 0-24 hours since admission) and at discharge (based on information from the 24 hours preceding discharge).
Suicide risk | Daily throughout the admission (range from 0 to about 150 days)
  Suicide risk is assessed daily throughout the admission by a clinical psychologist or psychiatrist treating the patient. It is scored using one item assessing if the patient has elevated risk of suicide using a binary scale (yes/no) and one item assessing if there is need for continuous observation of the patient to reduce suicide risk (yes/no).
Aggressive behavior | One score will be made 2 hours into each shift, a total of three times per day, every day, while the patient is admitted (range from 0 to about 150 days)
  Risk of aggressive behaviour are assessed three times per 24 hours by nurses using the Brøset Violence Checklist (BVC). The BVC is a 6-item scale assessing the presence of six observable behaviours on a binary scale (1=present/0=not present). The BVC has with good psychometric properties and the sum score (range 0-6) indicates risk of violence (low=0, moderate =1-2, high > 2).
Aggressive incidents | Aggressive incidents are not recorded at pre-specified time points, but the time and date are recorded if they occur throughout the duration of admission (range 0 to about 150 days).
  Actual incidents of aggressive behaviour will be systematically recorded using the Staff Observation Aggression Scale-Revised (SOAS-R) and interventions employed will be recorded by the nurses. The items in the SOAS-R specifies the context of the aggressive incident and the severity of the aggressive incident on a 0 to 100 scale (0 = not severe, 100 = very severe).
Medication use | Daily throughout the admission (range from 0 to about 150 days)
  Daily doses and classes of medications (e.g. antipsychotics, mood stabilizers, benzodiazepines, etc.) or other treatments or interventions prescribed per individual during admission will be recorded.
Admission status | Changes in admission status are not recorded at pre-specified times, but the time and date are recorded when they occur throughout the admission (range from 0 to about 150 days)
  If a patient is admitted involuntarily, the investigators will estimate the time until their status is reclassified as voluntary (as a marker of improved insight and mental capacity). Similarly change from voluntary to involuntary status and time to this reclassification will be recorded.
Patient Satisfaction and Benefit | At the day of discharge (range 0 to about 150 days)
  Mean levels of patient satisfaction with an admission are routinely assessed using the standard patient satisfaction questionnaire completed at discharge. The questionnaire was developed by Norwegian Institute of Public Health, is used throughout the Norwegian Health Care system and consists of 10 items scored on a 5-point Likert scale (1=low satisfaction). Some items are relevant to examining experiences of the different lighting conditions, (e.g. was the treatment was tailored to your situation?) Also, there are items related to side effects (see below). A specific item assesses the perceived benefit of the admission (1 = no benefit, 5 = very large benefit).
Side effects of the light environment | At the day of discharge (range 0 to about 150 days)
  The frequency of any side effects or adverse events experienced by individuals admitted to each lighting condition will be examined. The assessment comprises of the Headache and Eye Strain Scale (HES) supplement by additional items developed specifically for this trial and setting (and incorporated into the satisfaction questionnaire), 22 items in total. The HES assesses eight symptoms each of which is rated on a 4-point scale (ranging from absent = 0, to severe = 3) and is sensitive to exposure to different lighting conditions. Study participants are asked to rate any HES symptoms experienced during the course of admission and 14 further items that may represent side effects of acute psychiatric treatment (e.g. dizziness, gastro-intestinal disturbances, daytime sleepiness, poor sleep quality, and restlessness, etc.) that will also be rated using the same 4-point scale. Range of scores is 0 to 66 points.
Adverse effects of the light environment | Adverse effects are not recorded at pre specified times, but the time and date are recorded when they occur throughout the admission (range 0 to about 150 days)
  To capture any putative adverse events experienced during the admission the investigators will record any serious or untoward incidents (such as non-accidental and accidental deaths, near fatal events, severe violence, etc.). Also, the investigators will note if any patients are transferred out of the blue-depleted light environment because clinical opinion suggests that it may be having a detrimental effect on the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Kallestad, PhD, Principal Investigator — St. Olavs Hospital, Department of Research and Development
Locations (1):
- St. Olavs Hospital, Department Østmarka, Trondheim, Norway

REFERENCES:
- [Background] Scott J, Langsrud K, Vethe D, Kjorstad K, Vestergaard CL, Faaland P, Lydersen S, Vaaler A, Morken G, Torgersen T, Kallestad H. A pragmatic effectiveness randomized controlled trial of the duration of psychiatric hospitalization in a trans-diagnostic sample of patients with acute mental illness admitted to a ward with either blue-depleted evening lighting or normal lighting conditions. Trials. 2019 Aug 1;20(1):472. doi: 10.1186/s13063-019-3582-2. PMID 31370871
- [Derived] Kallestad H, Langsrud K, Simpson MR, Vestergaard CL, Vethe D, Kjorstad K, Faaland P, Lydersen S, Morken G, Ulsaker-Janke I, Saksvik SB, Scott J. Clinical benefits of modifying the evening light environment in an acute psychiatric unit: A single-centre, two-arm, parallel-group, pragmatic effectiveness randomised controlled trial. PLoS Med. 2024 Dec 6;21(12):e1004380. doi: 10.1371/journal.pmed.1004380. eCollection 2024 Dec. PMID 39642162

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03788993/SAP_000.pdf